CLINICAL TRIAL: NCT05195957
Title: Outcomes of Open Versus Robotic-assisted Laparoscopic Posterior Component Separation in Complex Abdominal Wall Repair A Retrospective Multicenter Case-control Study
Brief Title: Outcomes of Open Versus Robotic-assisted Laparoscopic Posterior Component Separation in Complex Abdominal Wall Repair
Acronym: EUROTAR
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Other Study IDs: 12/2021
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Wall Hernia
Keywords: Abdominal wall surgery; Open surgery; Robotic surgery; Transversus abdominis release; Posterior component separation technique
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rTAR: All consecutive patients undergoing bilateral robotic transversus abdominis release operation in the treatment of their ventral incisional hernia, are considered eligible for inclusion.
  Interventions: Procedure: Robotic tranversus abdominis release operation
- oTAR: All consecutive patients undergoing bilateral open transversus abdominis release operation in the treatment of their ventral incisional hernia, are considered eligible for inclusion.
  Interventions: Procedure: Open transversus abdominis release operation

INTERVENTIONS:
Procedure: Robotic tranversus abdominis release operation — Mini-invasive robotic-assisted TAR using either DaVinci Xi or Si systems and 6 laparoscopic ports.
  Groups: rTAR
Procedure: Open transversus abdominis release operation — Original open TAR using midline incision.
  Groups: oTAR

SUMMARY:
This is a retrospective European multicenter study evaluating surgical treatment of patients with a complex ventral incisional hernia using robotic-assisted laparoscopic transversus abdominis release (rTAR) or open transversus abdominis release (oTAR).

DETAILED DESCRIPTION:
Consecutive patients who undergo bilateral TAR in the treatment of their ventral incisional hernia in two European hernia centers are included in the study. A retrospective analysis of a prospectively maintained database and electronic patient files will be performed. Primary endpoint of the study was length of postoperative hospital stay. Secondary endpoints are intraoperative complications, in-hospital complications, overall and surgical site related complications during the first 30 postoperative days, overall and surgical site related complications during the reported follow-up period, and hernia recurrence during the reported follow-up period.

Data on the following variables wlll be collected.

* Patient characteristics: age, sex, body-mass index (BMI), comorbidities, smoking habits, previous hernia repair and hernia dimensions
* Intraoperatively: skin-to-skin operative time, wound contamination class (according to the center for disease control and prevention (CDC) classification)15, administration of antibiotics, mesh type used, mesh size, closure of the hernia defect, combined surgical procedures and intraoperative complications.
* Postoperatively at discharge: length of postoperative hospital stay and in-hospital complications.
* Postoperatively at 30 days after surgery: overall (according to the Clavien-Dindo classification)16 and surgical site related complications17, readmission rates during the first 30 days after surgery.
* During follow-up: duration of reported follow-up, reoperation rates and hernia recurrences during the reported follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing bilateral either open of robotic-assisted transversus abdominis release in the treatment of their ventral incisional hernia.

Exclusion Criteria:

* unilateral transversus abdominis release
* patients with a stoma or parastomal hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing bilateral either open of robotic-assisted transversus abdominis release in the treatment of their ventral incisional hernia.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | immediately after the surgery
  Postoperative treatment and follow-up period in hospital

SECONDARY OUTCOMES:
Complication rates | through study completion, an average of 1 year
  Postoperative complications during 30 days after surgery and longer follow-up
Recurrence and reoperation rates | through study completion, an average of 2 year
  Postoperative recurrence of hernia and possible reoperations for recurrence

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital Maria Middelares, Ghent, Belgium
- Tero Rautio, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes
All data is available for European Hernia Society researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After results are published without any time limitations
Access Criteria: When asked